CLINICAL TRIAL: NCT07025707
Title: Agreement and Reproducibility of Intraocular Lens Tilt and Decentration Measurements: A Comparison Between CASIA2 and CILT
Brief Title: Comparison of Two Different Methods for Calculating Intraocular Lens Tilt and Decentration
Status: Recruiting | Type: Observational
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0401-ST
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Intraocular Lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Agreement and Reproducibility of Intraocular Lens Tilt and Decentration Measurements: A Comparison between CASIA2 and CILT

DETAILED DESCRIPTION:
This prospective observational study evaluates the agreement and reproducibility of intraocular lens (IOL) tilt and decentration measurements obtained from two different imaging modalities: the CASIA2 anterior segment swept-source optical coherence tomography (AS-SS-OCT) system and the Calculator for Intraocular Lens Tilt (CILT) software, based on standardized anterior segment image analysis.

ELIGIBILITY:
Inclusion Criteria:

* planned cataract surgery
* agreement to participation

Exclusion Criteria:

* Zonulolysis
* Strabismus
* Reduced Compliance
* Axial length <20 or >25 mm
* Keratokonus
* PEX

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: planned cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular Lens Tilt (CASIA2 and CILT) | Measured during the pre-surgery examination under normal pupil conditions and after pharmacologic dilation (45 minutes post-mydriatic instillation).
  Intraocular lens (IOL) tilt, measured in degrees, assessed from anterior segment swept-source optical coherence tomography (AS-SS-OCT) images using the CASIA2 system and CILT software. Tilt is defined as the angle between the IOL plane and the corneal vertex.
Intraocular Decentration (CASIA2 and CILT) | Measured during the pre-surgery examination under normal pupil conditions and after pharmacologic dilation (45 minutes post-mydriatic instillation).
  Intraocular lens (IOL) decentration, measured in micrometers, assessed from anterior segment swept-source optical coherence tomography (AS-SS-OCT) images using the CASIA2 system and CILT software. Decentration is defined as the distance between the IOL center and the corneal vertex.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Amon, Prim. Univ. Prof. Dr., Study Chair — Hospital St. John of God
Locations (1):
- Krankenhaus der Barmherzigen Brüder Wien, Vienna, Vienna, Austria